CLINICAL TRIAL: NCT02543515
Title: Psychosocial and Clinical Characteristics Predicting Women's Acceptance of Office Hysteroscopy: An Observational Study
Brief Title: Psychosocial and Clinical Characteristics Predicting Women's Acceptance of Office Hysteroscopy
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar Tondela-Viseu (Other)
Collaborators: Marta Fernandes, M.D. MSc (Unknown); Sonia Gonçalves, M.D (Unknown); José Damasceno Costa, M.D. (Unknown); Antonio Pipa, M.D. (Unknown); Raquel Oliveira, MSc. (Unknown); nurse Catarina Mota (Unknown); nurse Carla Santos (Unknown)
Responsible Party: Principal Investigator, Antonio paulo, Consultant Obstetrician and Gynaecologist - Department of Obstetrics and Gynaecology, Hospital Centre Tondela-Viseu Assistant Professor Health Sciences Department, University of Aveiro - Portugal, Centro Hospitalar Tondela-Viseu
Other Study IDs: ASP/asp
Record Dates: First submitted 2015-08-29; First posted 2015-09-07 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Pelvic Girdle Pain
Keywords: following hysteroscopy
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: office hysteroscopy — diagnostic procedure
  Other Names: hysteroscopy,; mini-hysteroscopy

SUMMARY:
Study type:

Observational, prospective.

Objectives:

Primary:

Identify psychosocial and clinical factors that predispose to the occurrence of pain following office hysteroscopy

Secondary:

Stratify risk factors for pain previous Cesarean section and pain score repeat C section and pain score post-menopausal and pain score type of delivery and pain score body mass index and pain score history of dysmenorrhea and pain score, abnormal uterine bleeding and pain score previous surgery upon uterine cervix and pain score Characterize women's psychosocial profile and pain score Establish anxiety as a factor influencing pain perception using (State-Trait Anxiety Inventory for Adults).

Determine if there is a specified population who would benefit from procedure under anaesthesia

DETAILED DESCRIPTION:
Authors tend to compare pain in hysteroscopy in groups by scope size and variation in technique (e.g. 3mm versus 5mm scopes; vaginoscopic versus traditional speculum insertion approach), so score results reflect relative improvement in tolerability between groups, and they do not have as control an examination expected to be free of suffering.

To the investigators' knowledge there has to date never been an adequate judgement of the proportion of women in the group where pain is felt and should therefore be expected. Focus has always been put on the group of patients who are pain free (or where it is deemed acceptable).

Stating office hysteroscopy is painless because VAS score is halved by miniaturization seems an arbitrary statement for a small, but never the less important group of women.

It should be interesting to investigate factors which might contribute to pain in office hysteroscopy despite the fact the majority of the group will bear mild or no pain. The investigator believes that although reduction of scope size has brought about significant reduction in distress, it remains a painful procedure for some patients and therefore subjecting them to this ordeal may be regarded as an aggression; pain control interventions to reduce suffering might be considered (anxiolytic drugs, local, para-cervical or even general anaesthesia could be of interest in selected cases).

ELIGIBILITY:
Inclusion Criteria:

* women scheduled for office hysteroscopy Written informed consent; diagnosis of uterine abnormal bleeding, sonographic evidence of thickened endometrium, sterility workup, endometrial polyps or sub mucous myoma, foreign body extraction or insertion (i.e. sterilization) or other condition with indication for procedure and who meet study eligibility criteria; ability to fill in the study questionnaires.

Exclusion Criteria:

* refusal to participate in study innability to fill in the study questionnaires

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult women scheduled for office hysteroscopy.
  Eligibility criteria and informed consent:
  Written informed consent; diagnosis of uterine abnormal bleeding, sonographic evidence of thickened endometrium, sterility workup, endometrial polyps or sub mucous myoma, foreign body extraction or insertion (i.e. sterilization) or other condition with indication for procedure and who meet study eligibility criteria; ability to fill in the study questionnaires
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
office hysteroscopy in Nuligest | five to ten minutes after hystersocopy
  Pain score evaluated on a 10cm visual analogue scale
office hysteroscopy in parous women | five to ten minutes after hystersocopy
  Pain score evaluated on a 10cm visual analogue scale
office hysteroscopy in previous C section and repeat C section | five to ten minutes after hystersocopy
  Pain score evaluated on a 10cm visual analogue scale

SECONDARY OUTCOMES:
office hysteroscopy in post-menopausal women | five to ten minutes after hystersocopy
  Pain evaluated on a 10cm visual analogue scale
office hysteroscopy and body mass index | five to ten minutes after hystersocopy
  Pain evaluated on a 10cm visual analogue scale
office hysteroscopy and psychosocial profile (State-Trait Anxiety Inventory for Adults) | five to ten minutes after hystersocopy
  Pain evaluated on a 10cm visual analogue scale
Women's Satisfaction with office hysteroscopy according to pain perceived | five to ten minutes after hystersocopy
  Pain evaluated on a 10cm visual analogue scale and satisfaction questionnaires
office hysteroscopy in women with history of dysmenorrhea | five to ten minutes after hystersocopy
  Pain evaluated on a 10cm visual analogue scale
office hysteroscopy in women with abnormal uterine bleeding | five to ten minutes after hystersocopy
  Pain evaluated on a 10cm visual analogue scale
office hysteroscopy in women with previous surgery upon uterine cervix | five to ten minutes after hystersocopy
  Pain evaluated on a 10cm visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paulo, MD, Principal Investigator — Centro Hospitalar Tondela-Viseu
Locations (1):
- Centro Hospitalar Tondela Viseu, Viseu, Portugal